CLINICAL TRIAL: NCT02501239
Title: Health At Every Size and Acceptance and Commitment Therapy vs. Behavioral Weight Loss for Obesity and Depression in Women: A Randomized Controlled Trial
Brief Title: Health At Every Size and Acceptance and Commitment Therapy vs. Behavioral Weight Loss for Obesity and Depression in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Hitchcock Foundation (Other)
Responsible Party: Principal Investigator, Margit I. Berman, Associate Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D15151
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Depression; Obesity
MeSH Terms: conditions — Depression; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accept Yourself! Intervention (Experimental): Combined Health At Every Size and Acceptance and Commitment Therapy Psychotherapy Group
  Interventions: Behavioral: Accept Yourself!
- Behavioral Weight Loss (Active Comparator): Weight Watchers groups
  Interventions: Behavioral: Weight Watchers

INTERVENTIONS:
Behavioral: Accept Yourself!
  Other Names: HAES/ACT
  Arms: Accept Yourself! Intervention
Behavioral: Weight Watchers
  Arms: Behavioral Weight Loss

SUMMARY:
The primary aim of this project is to conduct a randomized controlled pilot study evaluating the feasibility and potential effectiveness of a newly developed combined Health At Every Size and Acceptance and Commitment Therapy (HAES/ACT) treatment, known as Accept Yourself! compared to a commercial behavioral weight loss program, Weight Watchers (WW). Obese women (BMI ≥ 30) with Major Depressive Disorder will be randomly assigned to one of these two treatments. Depression, physical health, and other psychosocial outcomes will be assessed prior to treatment, at post-treatment, and at 3, 6, 9, and 12-month follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Major Depressive Disorder (assessed using the Structured Clinical Interview for DSM-IV, SCID-IV)
* Body Mass Index (BMI) greater than or equal to 30
* Not taking medications or on stable medication regimens (i.e. no medication changes for six weeks prior to enrollment or during the study)

Exclusion Criteria:

* current substance dependence
* history of psychotic symptoms
* high risk of suicide/self-harm
* current enrollment in a weight-loss program
* weight loss surgery in the past year
* current psychotherapy
* inability to postpone weight loss or depression treatment interventions for the duration of the study
* taking antipsychotic, tricyclic, or oral corticosteroid medication
* unwilling to be randomized to the study treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2017-05-07 (Actual)

PRIMARY OUTCOMES:
Change in clinician assessed depression symptoms | At post-treatment (immediately following the three-month intervention) and at 3, 6, 9, and 12-month follow-up assessments.
  As assessed by clinician rated Hamilton Depression Rating Scale (HAM-D)
Change in self-reported depression symptoms | At post-treatment (immediately following the three-month intervention) and at 3, 6, 9, and 12-month follow-up assessments.
  As assessed by Patient Health Questionnaire-9 (PHQ-9)

SECONDARY OUTCOMES:
Change in fasting Lipids | At post-treatment (immediately following the three-month intervention) and at 12 month follow-up.
Change in systolic and diastolic blood pressure | At post-treatment (immediately following the three-month intervention) and 12 month follow up
Change in fasting blood glucose | At post-treatment (immediately following the three-month intervention) and 12 month follow up
Change in eating disorder symptoms, measured by the Eating Disorders Diagnostic Scale (EDDS) | At post-treatment (immediately following the three-month intervention) and at 3, 6, 9, and 12-month assessments.
Change in obesity-related quality of life, measured by the Obesity-Related Well-Being Questionnaire (ORWELL97) | At post-treatment (immediately following the three-month intervention) and at 3, 6, 9, and 12-month assessments.
Change in obesity stigma, measured by the Weight Self-Stigma Questionnaire (WSSQ) | At post-treatment (immediately following the three-month intervention) and at 3, 6, 9, and 12-month assessments.
Number of participants who did not complete an adequate dose of the intervention (at least 7 group visits) | At post-treatment (immediately following the three-month intervention)
Change in weight | At post-treatment (immediately following the three-month intervention) and 12 month follow up
  Note that we are assessing weight change primarily as a safety measure (i.e., to demonstrate no significant weight gain in intervention group).
Change in self-reported physical activity | At post-treatment (immediately following the three-month intervention) and at 12-month follow-up.
Change in cardiovascular fitness as assessed by six-minute walk test | At post-treatment (immediately following the three-month intervention) and at 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Margit I Berman, Ph.D, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Berman MI, Park J, Kragenbrink ME, Hegel MT. Accept Yourself! A Pilot Randomized Controlled Trial of a Self-Acceptance-Based Treatment for Large-Bodied Women With Depression. Behav Ther. 2022 Sep;53(5):913-926. doi: 10.1016/j.beth.2022.03.002. Epub 2022 Mar 23. PMID 35987548